CLINICAL TRIAL: NCT00978666
Title: Neural Dysfunction of Interoception in Adolescents Diagnosed With Anorexia Nervosa
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Imaging Study in Adolescents With Anorexia Nervosa
Acronym: ADOL_AN
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amanda Grethe, Principal Investigator, University of California, San Diego
Other Study IDs: 090008; R21MH086017 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-17 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy controls: Healthy comparison adolescent females
- Anorexia Nervosa: Adolescent females currently ill with Anorexia Nervosa, restricting type

SUMMARY:
The purpose of this study is to use fMRI imaging technology to examine areas in the brain related to appetite, reward and cognition in adolescent women with eating disorders as compared to those who have never had an eating disorder. Better understanding biologic vulnerabilities in women with anorexia is essential for developing more effective treatment options.

DETAILED DESCRIPTION:
Individuals with anorexia nervosa (AN) have aberrant feeding behavior, disturbances of emotionality and impulse control, and have high rates of relapse after weight restoration (Carter et al., 2004; Halmi et al., 2003). There is no proven treatment that reverses symptoms. Although imaging studies in individuals recovered from AN (REC AN) suggest that these symptoms are related to dysfunction of the striatal, insular, and prefrontal areas, less is known about the biology of these core symptoms in currently ill individuals (ILL AN). This application will use blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (fMRI) to examine neural substrates underlying appetitive, reward, and cognitive dysregulation in ill AN. We will study 22 adolescent women currently ill with AN and 22 healthy adolescent control women (CW), all of whom are 14 to 18 years old.

The specific aims of the project are:

AIM 1: The anterior insula (AI), orbitofrontal cortex (OFC), and associated regions integrate sensory/hedonic aspects of taste and interoceptive awareness in the service of homeostasis. We hypothesize that restricted eating and weight loss occur in AN because a palatable food elicits little reward.

AIM 2: Little in life is rewarding to individuals with AN aside from weight loss, and they tend to be overconcerned with future consequences. We predict that ill AN will show an inability to discriminate positive and negative feedback reflecting aberrant anterior ventral striatum (AVS) limbic function.

AIM 3: AN tend to be rigid, inflexible and behaviorally inhibited. We will use a stop task (Band et al., 2003; Logan et al., 1984; Matthews et al., 2005) to characterize the neural substrates of inhibitory motor control. We hypothesize that ill AN, relative to CW, will show a demand-specific alteration of a fronto-subthalamic circuit that is necessary for motor inhibition (Aron et al., 2004).

AIM 4: In an exploratory aim, we propose to examine how clinical, cognitive, and personality/temperament measures might be correlated to either the BOLD response and/or the integrity of frontostriatal connectivity as determined using diffusion tensor imaging (DTI).

Taken together, these aims will enable us to better characterize cognitive and limbic dysfunction in these populations. Understanding biologic vulnerabilities in AN is critical for developing effective treatment interventions for this often chronic and deadly disorder. In addition, there is a lack of understanding of appropriate methodologies necessary to address the unique problems inherent in the study of ill AN. Thus, this project will also characterize confounding factors, such as brain volume, energy metabolism, development stages, and gonadal steroids, with the intent that a future project will incorporate the methodology needed to rigorously investigate this population.

ELIGIBILITY:
Participants w/ Anorexia Inclusion Criteria

* Female
* Ages 12-18
* Right Handed
* Active AN diagnosis (within last 6 months), excluding amenorrhea criteria
* IBW 70-87% Exclusion Criteria
* Male
* Left Handed
* Does not meet AN criteria within last 6 months
* Alcohol/drug dependence in the 3 months prior to study
* Alcohol/drug use within the 30 days prior to scan. Tox Screen will be administered at GCRC.
* Use of antipsychotic medication in 3 months prior to study (SSRI OK)
* Current diagnosis of severe major effective d/o or anxiety d/o or other psychopathology that might interfere with ability to participate e.g requiring inpatient hospitalization or medication
* Pregnancy or lactation
* Organic brain syndromes, dementia, psychotic disorders or mental retardation
* Neurological or medical disorders such as seizure disorder, renal disease including pyelonephritis and chronic cystitis, impaired renal function including hyponatremia (less than 135meq/l), hypokalemia, raised BUN (more than 15mg/dl), diabetes, thyroid disease (hypo and hyper), EKG indicative of electrolyte imbalance
* Lack of effective birth control during 15 days before the scan. A Urine pregnancy test will be conducted within 24 hours of the scan
* Insufficient English

Healthy Volunteer Participants Inclusion criteria

* Female
* Ages 12-18
* Right Handed
* IBW between 90% and 120% Exclusion Criteria
* Male
* Left Handed
* Current or past psychiatric (definitive Axis I) disorder
* Alcohol/drug use within the 30 days prior to scan
* Pregnancy or lactation
* Organic brain syndromes, dementia, psychotic disorders or mental retardation
* Neurological or medical illness as indicated by lab tests, medical and psychiatric histories and physical examination
* Any stigmata suggestive of eating disorder
* Any first degree relatives with an Eating Disorder
* Any first degree relative with a current/past major psychiatric disorder (depression and alcoholism taken on a case by case basis and measured by severity)
* Insufficient English

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants with anorexia nervosa will be selected from the community as well as from local medical clinics and eating disorder treatment centers. Healthy volunteers will be selected from the community at large.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCSD Eating Disorder Treatment and Research Program, La Jolla, California, United States

REFERENCES:
- See also: Related Info — http://eatingdisorders.ucsd.edu/